CLINICAL TRIAL: NCT05464225
Title: Colorado Oral Strengthening Device
Acronym: COSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Davis Phinney Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-1850
Record Dates: First submitted 2022-07-14; First posted 2022-07-19 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: tongue strength; novel exercise
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Prospective cohort of 60 individuals with Parkinson's will be randomly assigned (please read 'Participant Randomization' below) to either exercise using the COSD or to standard of care using tongue depressors, as per the request of the funding source.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COSD (Experimental): Participants assigned to the COSD, will use the investigational device.
  Interventions: Device: COSD
- SOC (Active Comparator): Tongue depressors are the standard-of-care so the control group will use these instead of the investigational "Colorado Oral Strengthening Device."
  Interventions: Device: SOC

INTERVENTIONS:
Device: COSD — The exercise protocol will include using the tongue to compress the COSD against the hard palate, or against the tongue depressor for 30 repetitions, 3 times per day, on 3 days of the 7-day week. For the first week, the participants who are in the COSD group will be issued a COSD bulb that corresponds to no less than 60% of their baseline maximum strength. After week 1, they will switch to a COSD bulb that corresponds to no less than 80% of their maximum tongue strength for the remaining 7 weeks.
  Arms: COSD
Device: SOC — The exercise protocol will include using the tongue to compress the COSD against the hard palate, or against the tongue depressor for 30 repetitions, 3 times per day, on 3 days of the 7-day week. For the tongue depressor group, they will be given 8 tongue depressors, which are disposable, for the duration of the study.
  Other Names: Tongue Depressor
  Arms: SOC

SUMMARY:
University of Colorado is looking for adults with Parkinson's disease to participate in a research study. The study aims to explore how a novel low technology device can achieve an increase in tongue strength comparable to standard of care exercise using tongue depressors but with the kinematics and simple biofeedback of existing high cost devices. Research has shown that tongue resistance exercises paired with biofeedback have resulted in improved tongue strength to support chewing, control of food and liquid in the mouth, and propulsion of material for a swallow.

DETAILED DESCRIPTION:
When an individual contacts the PI or the department research coordinator, a preliminary screen will be administered for any obvious exclusion. If there are no exclusions, the first visit will be scheduled. At this initial visit, a full description of the study and exercise protocol will be provided. A health history questionnaire and an EAT-10 questionnaire will be administered.

If consent is obtained, baseline tongue strength will be measured using the IOPI device. Individuals with Parkinson's will be randomized to exercise with the COSD or with the tongue depressors. Those who will use the COSD will be start with no less than 60% max strength and receive an exercise log. Those using the tongue depressors will also receive an exercise log.

All participants will receive a full demonstration of the exercise and will be asked to return the demonstration.

The second visit will be scheduled for all participants the following week. At that time, the EAT-10 and tongue strength will be re-assessed. The exercise logs will be reviewed to ensure compliance. Participants using the COSD will be issued a new device that is no less than 80% of their max strength.

The third visit will be scheduled the following week (week 3). The EAT-10 questionnaire and tongue strength will be reassessed. The exercise log will be reviewed for compliance. COSD will be inspected for any signs of wear and a new one will be issued if the device appears worn.

The last 2 visits will be scheduled during weeks 6 and 8 of the exercise protocol. The EAT-10 and tongue strength will be re-assessed, and the exercise log will be reviewed for compliance. The COSD will be inspected for any signs of wear and a new one will be issued if the device appears worn. In addition, during the final visit, all participants will be asked to complete a questionnaire regarding their satisfaction with the exercise device they were assigned. The COSD will be collected at that visit.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 89 years old(inclusive)
2. Diagnosis of Parkinson's Disease
3. Hoen and Yahr stage II-IV
4. Signs or symptoms of dysphagia evidenced by an EAT-10 score of 3 or more

Exclusion Criteria:

1. Unwilling to sign the informed consent
2. Atypical Parkinson's Disease, Parkinson Plus, Lewy Body Dementia, Multiple System Atrophy
3. History of head or neck cancer
4. History of seizures
5. Current or past disorders of the jaw
6. Allergy to device materials

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Change in Tongue Strength, as measured in kPa via IOPI | Baseline, up to 8 weeks.
  Tongue Strength, as measured in kPa via IOPI with measurements that are equal to or higher compared to baseline at follow-up visits at weeks 2,3,6 and 8 from initial visit. Tongue strength will be assessed using The Iowa Oral Pressure Instrument (IOPI). IOPI measures tongue strength with max pressure (kPa) ranging from 0 to 110 with an average of 50-60 kPa depending on age. Higher kPa is associated with increased tongue strength.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Cuadrado, Principal Investigator — Department of Otolaryngology
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No